CLINICAL TRIAL: NCT00191568
Title: A Phase II Trial of Adjuvant Treatment With Gemcitabine and Oxaliplatin Followed by Concomitant Gemcitabine and Radiation Therapy in Patients With Resected Pancreatic Adenocarcinoma
Brief Title: Gemcitabine, Oxaliplatin and Radiotherapy in Treating Patients With Completely Resected Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6866; B9E-MC-S298
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin; Radiotherapy

INTERVENTIONS:
Drug: Gemcitabine
Drug: Oxaliplatin
Procedure: Radiotherapy

SUMMARY:
A non-randomized phase II study to determine the efficacy and safety of the combination of Gemcitabine and Oxaliplatin followed by Gemcitabine and radiotherapy in patients with surgically resected pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the pancreas
* Patient have undergone a potentially curative resection
* No previous irradiation to the planned field
* Negative pregnancy test for child bearing women

Exclusion Criteria:

* Non-adenocarcinoma pancreatic cancer
* Treatment with any drug within the last 30 days that has not received regulatory approval.
* Serious systemic disorder
* Metastatic disease
* Pregnancy, breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2002-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To evaluate recurrence free one year survival, time to disease progression and local recurrence rate, analyzed at the end of the study

SECONDARY OUTCOMES:
To assess overall survival at the end of the 24 months follow up period;To assess acute and late toxicity (every month for the first 3 months and then every three months for 24 months after treatment discontinuation)

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- France (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) MON-FRI 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Grenoble
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) MON-FRI 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) MON-FRI 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) MON-FRI 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) MON-FRI 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) MON-FRI 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Pierre-Bénite

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com